CLINICAL TRIAL: NCT03703609
Title: Effects of Tele-yoga on Physical Function, Health-related Quality of Life, Symptoms of Anxiety and Depression in Long-term Conditions
Brief Title: Effects of Tele-yoga in Long-term Conditions
Acronym: TELEYOGA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Anna Stroemberg, professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2017/225-31
Record Dates: First submitted 2018-10-07; First posted 2018-10-12 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Chronic Disease
Keywords: yoga; rehabilitation; physical activity; quality of life; anxiety; depression
MeSH Terms: conditions — Chronic Disease; Motor Activity; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: The study is a single-blind parallel two-arm randomized controlled study with 1:1 distribution to intervention and control group. In total 300 persons with long-term conditions will be recruited from three hospitals and randomized to an intervention of medical yoga at home (tele-yoga) using a live videoconference link and a yoga-app on the participants tablet for 12 weeks or a control group receiving individual advice of physical activity. Data will be collected at baseline measurement, after 3 and 6 months.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Analyst blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-yoga (Experimental): Intervention of doing medical yoga at home (tele-yoga) using (1) an online videoconference system (zoom) for particpating in group-yogaled by a live yoga instructor for 60 minutes twice a week and (2) daily individual yoga for a minimum of 10 minutes using a yoga-app. Participants are provided with a tablet with conference system zoom and yoga app for 12 weeks
  Interventions: Behavioral: Tele-yoga
- Individual physical activty advice (No Intervention): The active control group will receive advice to be physically active that corresponds to the intervention group in time and effort, equivalent to 60 minutes for 2 days a week and a minimum of 10 minutes for 5 days a week. To compensate for the extra attention received by the intervention group by the instructor via tele-yoga group, the participants in the activecontrol group's patients will be dialed or have SMS contact (the participant chooses a type of contact) with a physiotherapist or nurse after 2, 4, 8 and 12 weeks.

INTERVENTIONS:
Behavioral: Tele-yoga — Participants will get a 60 min tele-yoga session biweekly led by a certified medical yoga instructor via live videoconference link on the participants tablet. Each participant will perform a total of 20-24 yoga instructor-led sessions over a 12-week period. A session will contain 10 min breathing exercises, 40 min of yoga and 10 min relaxation/meditation. Before and at the end of each session, participants can discuss their experiences or ask questions to the instructor online. The tablet also includes an app with instructions (text, pictures, and sound files) for yoga positions, breathing and meditation. Participants are encouraged to practice yoga at home individually with one goal of one session a day for a minimum of 10 minutes.
  Arms: Tele-yoga

SUMMARY:
Long-term illness is common in the Swedish population, especially among older people. These conditions are often associated with impaired quality of life due to high physical and psychological symptom-burden. Medical Yoga is a therapeutic form of Kundalini Yoga with simple movements, breathing exercises and meditation. For people with serious long-term illness, it can be difficult to attend regular yoga-classes. In this study, the investigators therefore set out to develop a tele-yoga intervention and evaluate the impact of medical yoga remotely at home with regard to physical function, quality of life, symptoms of anxiety and depression, biomarkers, sleep and cognition in people with long-term conditions. Health care utilisation as well as satisfaction and experiences with the exercise form and technology used will also be assessed. The evaluation will be conducted in 150 people with long-term illness recruited from three hospitals (one university hospital and two county hospital) randomised to receive either an intervention with medical yoga remotely at home (tele-yoga) for 12 weeks or a control group receiving individualised training to the same extent. The tele-yoga intervention will be provided remotely in the home via a video-transferred yoga instructor twice a week using a tablet and an app for individual daily exercise. Data will be collected at baseline, after 3 and 6 months.

Despite evidence that physical activity improves quality of life and functional capacity and probably survival, it is difficult to motivate and enable elderly people with long-term conditions to engage in physical and mental rehabilitation. In this study, we will test whether a new method conveyed through a technical solution remotely can increase patients' activity and well-being through allowing tele-yoga at home. Can health care resources be reduced, financial gains can also be made.

The study aims to evaluate the impact of medical yoga remotely at home with regard to physical function, quality of life, symptoms of anxiety and depression, biomarkers, sleep and cognition in people with long-term conditions. The investigators will also measure health care utilisation as well as satisfaction and experiences with the exercise form and technology used. The evaluation will be conducted in 300 people with long-term illness randomised to either tele-yoga or a control group.

DETAILED DESCRIPTION:
A sub-study will be conducted exploring physiological effects of yoga in participants with heart failure. The sub-study will include 40 of the patients with heart failure included in the main study. In the sub-study six additional measures will be performed at baseline and after 3 months in 20 study participants with heart failure in the intervention group; ergospirometry, echocardiography, Holter ECG, microcirculation using the epos system, maximal inspiratory and expiratory pressure. There will be four additional measures in 20 participants from the control-group at baseline and after 3 months; Holter ECG, microcirculation using the epos system and maximal inspiratory and expiratory pressure.

ELIGIBILITY:
Inclusion Criteria:

* Long-term illness and cared for at the cardiology clinic or intensive care clinic for at least 48 hours in the last 3-36 months.
* Clinically stable condition at the inclusion.

Exclusion Criteria:

* Inability to fill in questionnaires.
* Inability to participate in the intervention.
* Expected survival of less than 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Composite end-point including physical fuction, health-related quality of life and symptoms of anxiety and depression. | 3 months
  The composite weighed score consists of physical ability (6 min walking test), Health-realted quality of Life (EQ-5D) and symptom of anxiety and depression (HADS). Based on the change in these 3 variables, a patient can get a score between -3 and + 3 based on the increase, decrease or no change in 6 min walk test, HADS, and EQ5D. The weighted variable will be categorised as improved, deteriorated or unchanged after 3 months.

SECONDARY OUTCOMES:
Aerobic capacity/endurance | 3 and 6 months
  6 min walk test is a sub-maximal exercise test used to assess aerobic capacity and endurance. Measures the distance in meters covered over a time of 6 minutes
Symptoms of Anxiety and Depression | 3 and 6 months
  Hospital anxiety and depression scale is a 14 item scale that generates ordinal data 0-3. Seven of the items relate to anxiety, range 0-21 and seven relate to depression, range 0-21.
Health-related quality of life | 3 and 6 months
  The EQ-5D comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The responses generate ordinal data from 1-5 for each dimension. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale 0-100 mm, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'.
Physical activity | 3 and 6 months
  Actigraph
Cognition | 3 and 6 months
  Montreal Cognitive Assessment including short-term memory, visual abilities, executive functions, attention, concentration, working memory, language and orientation to time and place. Scores range between 0 and 30. A score of 26 or over is considered to be normal.
Sleep | 3 and 6 months
  Minimal insomnia symptom scale is a sleep questionnaire with 3 items that generates ordinal data. Range 0-12.
Exercise Motivation | 3 and 6 months
  The Exercise Motivation Index includes 15 items that generates ordinal data on the motives of participating in physical exercise. Range 0-60.
Lower body strength | 3 and 6 months
  Sit to stand test measure the number of uprising from a chair during 30 seconds.
Gait speed | 3 and 6 months
  Gait speed test meaures the time it takes in seconds to walk 10 meter at self-selected pace.
Health Health | 3 and 6 months
  One general health question from RAND 36 genreating an ordinal data response from 1 (poor health)-5 (excellent health).
Life satisfaction | 3 and 6 months
  Cantril ladder of Life is a measurement technique that asks people to rate their present, past, and anticipated future satisfaction with life on a scale anchored by their own identified values from 1 to 10.

OTHER OUTCOMES:
HcCRP | 3 and 6 months
  High sensitivity C-reactive protein (CRP) will be used as a routine marker of inflammation. Blood samples were collected while the patients were at rest in a supine position using EDTA-vials. The vials were chilled on ice before centrifugation at 3000 g, 4oC and then frozen at -70ºC. No sample was thawed more than twice. CRP was analysed using latex-enhanced turbidimetric immunoassay (Roche Diagnostics GmbH, Vienna, Austria) with a lower detection limit of 0.03 mg/L and coefficient of variation of 1.7%.
Cost-effectiveness | 6 months
  Health care utilisation through medical charts/registries. The cost of the intervention will also be calculated.
Adherence | 3 months
  The adherence will be measured through attendance in video groups and the use of yoga app The minutes each participant have used to perform individual yoga training will be measured via a statistical software incorporated in the yoga app.
Qualitative interviews | 3 months
  Telephone interviews about yoga, tele-yoga, user-friendliness and use of technology in the tele-yoga group
Quality-adjusted life-year (QALY) | 6 months
  Will be obtained from the EQ-5D

CONTACTS AND LOCATIONS:
Overall Officials: Anna Stromberg, PhD, Principal Investigator — Linkoeping University
Locations (4):
- Sweden (4):
  - Mälardals hospital, Eskilstuna
  - Ryhov hospital, Jönköping
  - Linköpings University hospital, Linköping
  - Vrinnevi Hospital, Norrköping

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hedbom T, Liljeroos M, Thylen I, Orwelius L, Jaarsma T, Stromberg A. Expectations of Tele-Yoga in Persons With Long-Term Illness: Qualitative Content Analysis. J Med Internet Res. 2023 Sep 13;25:e36808. doi: 10.2196/36808. PMID 37703082
- See also: Study website — https://liu.se/forskning/teleyoga-nar-ost-moter-vast